CLINICAL TRIAL: NCT03126591
Title: An Open-Label, Multicenter, Phase 1a/1b Study of Olaratumab (LY3012207) Plus Pembrolizumab (MK3475) in Patients With Unresectable Locally Advanced or Metastatic Soft Tissue Sarcoma (STS) Who Have Failed Standard Treatments
Brief Title: A Study of Olaratumab (LY3012207) Plus Pembrolizumab in Participants With Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15847; I5B-MC-JGDQ (Other: Eli Lilly and Company); 2016-001949-19 (EudraCT Number); KEYNOTE-505 (Other: Merck Sharp & Dohme, LLC); MK-3475-505 (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 15 milligrams per kilogram (mg/kg) Olaratumab + 200 milligrams (mg) Pembrolizumab - Dose Escalation (Experimental): Participants received15 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
  Interventions: Drug: Olaratumab; Drug: Pembrolizumab (KEYTRUDA®)
- 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation (Experimental): Participants received 20 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
  Interventions: Drug: Olaratumab; Drug: Pembrolizumab (KEYTRUDA®)
- 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion (Experimental): Participants received 20 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
  Interventions: Drug: Olaratumab; Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207
Drug: Pembrolizumab (KEYTRUDA®) — Administered IV
  Other Names: MK3475

SUMMARY:
The purpose of this study is to evaluate the safety of olaratumab plus pembrolizumab in participants with previously treated advanced or metastatic soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced unresectable or metastatic STS, not amenable to curative treatment and after available standard therapies have failed to provide clinical benefit. Note: Participants with a diagnosis of Grade 1 liposarcoma (atypical lipomatous neoplasms) are eligible if there is histological or radiographic evidence of evolution to more aggressive disease.
* Presence of measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Must be able to provide tumor tissue obtained within 6 months of study enrollment. If such tissue is not available, a newly obtained core or excisional biopsy of a tumor lesion must be performed.
* Have an anticipated life expectancy of ≥3 months.

Exclusion Criteria:

* Have received any previous systemic therapy (including investigational agents) targeting PD-1/programmed cell death ligand 1 (PDL-1) or PD-1/PDL-2 signaling pathways (including previous participation in Merck MK-3475 trials). Prior treatment with olaratumab is allowed. Prior therapy with other immune checkpoint inhibitors, including but not limited to, anti-CD137 antibody or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody, is not permitted.
* Have known active central nervous system (CNS) metastasis and/or carcinomatous meningitis. Participants with treated CNS metastases are eligible for this study if they have not received corticosteroids and/or anticonvulsants within 7 days of study treatment, and their disease is asymptomatic and radiographically stable for at least 60 days.
* Have active autoimmune disease or other syndrome that requires systemic steroids or autoimmune agents in the past 2 years.
* History of interstitial lung disease or non-infectious pneumonia.
* Have received a live-virus vaccine within 30 days prior to planned treatment start.
* Have histologically or cytologically confirmed Kaposi's sarcoma or gastrointestinal stromal tumor (GIST).
* Have inflammatory bowel disease for which the participant has used immunosuppressive agents within the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium
- Herlev and Gentofte Hospital, Herlev, Denmark
- Gustave Roussy, Villejuif, France

REFERENCES:
- See also: A Study of Olaratumab (LY3012207) Plus Pembrolizumab in Participants With Advanced or Metastatic Soft Tissue Sarcoma — https://trials.lilly.com/en-US/find/completed?trialname=%20I5B-MC-JGDQ&externalRequestID=68cbce79-fbf1-46c5-852a-338ca6e2be85

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the study were considered a completer.
Groups:
- 15 Milligrams/Kilogram (mg/kg) Olaratumab + 200 Milligrams (mg) Pembrolizumab - Dose Escalation: Participants received15 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
Period: Overall Study
Arm/Group | 15 Milligrams/Kilogram (mg/kg) Olaratumab + 200 Milligrams (mg) Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Started | 7 | 6 | 28
Received at Least 1 Dose of Study Drug | 7 | 6 | 28
Completed | 0 | 0 | 1
Not Completed | 7 | 6 | 27
Not completed — Death | 6 | 3 | 17
Not completed — Progressive Disease | 0 | 1 | 2
Not completed — Terminated by Sponsor | 0 | 1 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation: Participants received15 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
- 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion: Participants received 20 mg/kg Olaratumab administered IV on Day 1 and Day 8 in addition to 200 mg Pembrolizumab administered IV on Day 1 of a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion | Total
Number analyzed (Participants) | 7 | 6 | 28 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.57 (14.97) | 56.00 (14.31) | 57.82 (12.71) | 56.83 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 17 | 26
  Male | 2 | 2 | 11 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 7 | 3 | 21 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 2 | 5 | 10
  United States | 4 | 2 | 14 | 20
  Denmark | 0 | 0 | 4 | 4
  France | 0 | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Olaratumab Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event (AE) during Cycle 1 that is possibly related to the study drug and fulfills any 1 of the following criteria using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0:
  * Grade ≥3 nonhematologic toxicity, with exceptions
  * Grade 4 anemia
  * Grade 4 neutropenia or leukopenia of >5 days duration
  * Febrile neutropenia
  * Grade 3 thrombocytopenia with clinically significant bleeding or Grade 4 thrombocytopenia
  * Any other significant toxicity deemed to be dose limiting
Time Frame: Cycle 1 (21 Days)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
participants | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Olaratumab
Description: Maximum observed serum concentration of Olaratumab
Time Frame: Cycle 1 and Cycle 3 Day (D) 1: Predose, 1, 2, 5, 24, 96, 168 hours Postdose; Cycle 1 and Cycle 3 Day 8: Predose, 1, 2, 5, 48, 168, 336 hours Postdose
Population: All enrolled participants who received at least 1 dose of study drug and have at least 1 post-baseline evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 6 | 5 | 28
μg/mL
  C1D1 | 385 (19) | 548 (16) | 529 (19)
  C1D8: number analyzed (Participants) | 2 | 5 | 26
  C1D8 | NA (NA) — Individual values reported: 710 μg/mL and 472 μg/mL | 682 (17) | 693 (24)
  C3D1: number analyzed (Participants) | 1 | 4 | 17
  C3D1 | NA (NA) — Individual value reported: 694 μg/mL | 703 (14) | 761 (34)
  C3D8: number analyzed (Participants) | 1 | 5 | 18
  C3D8 | NA (NA) — Individual value reported: 819 μg/mL | 855 (8) | 845 (34)

3. Secondary Outcome: PK: Minimum Serum Concentration (Cmin) of Olaratumab
Description: Cmin was the concentration of olaratumab in the sample taken just prior to the following dose.
Time Frame: Cycle 1 and Cycle 3 Day 1: Predose, 1, 2, 5, 24, 96, 168 hours Postdose; Cycle 1 and Cycle 3 Day 8: Predose, 1, 2, 5, 48, 168, 336 hours Postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 24
μg/mL
  C1D1: number analyzed (Participants) | 7 | 5 | 24
  C1D1 | 129 (20) | 141 (13) | 135 (35)
  C1D8: number analyzed (Participants) | 5 | 6 | 24
  C1D8 | 132 (38) | 144 (35) | 134 (59)
  C3D1: number analyzed (Participants) | 3 | 5 | 18
  C3D1 | 272 (38) | 320 (17) | 263 (62)
  C3D8: number analyzed (Participants) | 2 | 5 | 17
  C3D8 | NA (NA) — Individual values reported: 212 μg/mL and 350 μg/mL | 207 (45) | 190 (79)

4. Secondary Outcome: PK: Elimination Half-Life (t½) of Olaratumab
Description: Terminal elimination half-life of Olaratumab
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 6 | 5 | 27
days
  C1D1: number analyzed (Participants) | 6 | 4 | 27
  C1D1 | 5.20 (40) | 4.47 (15) | 4.12 (22)
  C1D8: number analyzed (Participants) | 2 | 5 | 24
  C1D8 | NA (NA) — Individual values reported: 9.70 days and 8.94 days | 7.82 (13) | 7.53 (34)
  C3D1: number analyzed (Participants) | 1 | 4 | 16
  C3D1 | NA (NA) — Individual value reported: 9.71 days | 6.40 (24) | 6.39 (73)
  C3D8: number analyzed (Participants) | 1 | 5 | 13
  C3D8 | NA (NA) — Individual value reported: 15.2 days | 9.42 (29) | 8.84 (51)

5. Secondary Outcome: Number of Participants With Anti-Olaratumab Antibodies (ADA) When Administered in Combination With Pembrolizumab
Description: Detection of ADA in the presence of Olaratumab
Time Frame: Predose Cycle 1 Day 1 through Follow Up (up to 6 months)
Population: All enrolled participants who received at least one dose of study drug and had at least one anti-olaratumab antibody positive result.
Measure: Number; unit: participants
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
participants | 1 | 1 | 2

6. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: ORR was defined as the percentage of participants who achieved a CR or PR out of all participants treated, measured and recorded by Response Evaluation Criteria in Solid Tumors (RECIST v1.1). CR was defined as the disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm; tumor marker results must have normalized. PR was defined as at least a 30% decrease in the sum diameter of target lesions (taking as reference the baseline sum diameters). Long term follow up began the day after the safety follow up period was completed.
Time Frame: Baseline to Measured Progressive Disease (PD) or Start of New Anti-Cancer Therapy (up to 28 months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
percentage of participants | 0 [NA to NA] — 95% Confidence Interval could not be calculated as zero participants attained the event. | 0 [NA to NA] — 95% Confidence Interval could not be calculated as zero participants attained the event. | 21.4 [6.2 to 36.6]

7. Secondary Outcome: Disease Control Rate (DCR): Percentage of Participants With a Best Response of CR, PR or Stable Disease (SD)
Description: DCR was defined according to RECIST v1.1 as the percentage of participants who have achieved CR, PR or stable disease (SD). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Long term follow up began the day after the safety follow up period was completed.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (up to 28 months)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
percentage of participants | 14.3 [0.0 to 40.2] | 66.7 [28.9 to 100.0] | 53.6 [35.1 to 72.0]

8. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined according to RECIST v1.1 as the time from the date of the first CR or PR to the first date of PD or death from any cause, whichever is earlier. For each participant who was not known to have died or to have had a progression of disease as of the data inclusion cut-off date, DOR was censored at the date of last objective response assessment prior to the date of any subsequent systemic anticancer therapy. Long term follow up began the day after the safety follow up period was completed.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (up to 24 months)
Population: All enrolled participants who received at least one dose of study drug and who had a PR or CR. Number of participants censored in 20 mg/kg Dose Expansion arm = 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 0 | 0 | 6
months |  |  | 16.16 [1.68 to NA] — There were not enough events to estimate the upper confidence limit.

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) time was defined as the time from the date of start of study treatment to the first date of PD (symptomatic or objective) or death due to any cause, whichever occurs first. For participants who were not known to have died or progressed as of the data-inclusion cut-off date, PFS time was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systemic anticancer therapy. Long term follow up began the day after the safety follow up period was completed.
Time Frame: Baseline to Measured Progressive Disease or Death Due to Any Cause (up to 28 months)
Population: All enrolled participants who received at least one dose of study drug. Number of participants censored per arm: 15 mg/kg Olaratumab - Dose Escalation = 2 participants; 20 mg/kg Olaratumab - Dose Escalation = 0 participants; 20 mg/kg Olaratumab - Dose Expansion = 5 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
months | 1.38 [1.28 to NA] — There were not enough events to estimate the upper confidence limit. | 2.71 [1.38 to NA] — There were not enough events to estimate the upper confidence limit. | 2.69 [1.31 to 4.07]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. Data was censored for any participant who was not known to have died or was lost to follow up. Long term follow up began the day after the safety follow up period was completed.
Time Frame: Baseline to Death from Any Cause (up to 35 months)
Population: All enrolled participants who received at least one dose of study drug. Number of participants censored per arm: 15 mg/kg Olaratumab - Dose Escalation = 1 participant; 20 mg/kg Olaratumab - Dose Escalation = 3 participants; 20 mg/kg Olaratumab - Dose Expansion = 12 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
Number analyzed (Participants) | 7 | 6 | 28
months | 11.37 [5.62 to NA] — There were not enough events to estimate the upper confidence limit. | 16.39 [6.01 to NA] — There were not enough events to estimate the upper confidence limit. | 14.78 [12.58 to NA] — There were not enough events to estimate the upper confidence limit.

ADVERSE EVENTS:
Time Frame: Baseline through completion of safety follow up period (up to 35 months)
Description: All enrolled participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly. The safety follow-up period began one day after the participant was no longer continuing treatment and lasted up to 90 days.
Arm/Group | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion
All-Cause Mortality (participants affected / at risk) | 6/7 | 3/6 | 17/28
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/6 | 15/28
Other Adverse Events (participants affected / at risk) | 7/7 | 5/6 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation (N=7) | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation (N=6) | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 15 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation (N=7) | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Escalation (N=6) | 20 mg/kg Olaratumab + 200 mg Pembrolizumab - Dose Expansion (N=28)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 7 (16)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 9 (11)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3) | 11 (15)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (3)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Cystoscopy (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 2 (4) | 0 (0) | 3 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3) | 4 (8)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 5 (17)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (6)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 3 (10)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 6 (7)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0/2 (0) | 0/2 (0) | 1/11 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 7 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03126591/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03126591/SAP_001.pdf